CLINICAL TRIAL: NCT03920579
Title: A Sequence-randomized, Open-label, 3-way Crossover, Single Oral Dose Clinical Trial to Investigate the Pharmacokinetic Characteristics and Safety/Tolerability According to Formulations of CKD-386 in Healthy Male Volunteers
Brief Title: A Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of CKD-386 in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 183PK18034
Record Dates: First submitted 2019-04-08; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Hypertension; Dyslipidemias
Keywords: CKD-386; Pharmacokinetics; D326; D337; D013
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: CKD-386 formulation 1(1 tab, once) / Period 2: CKD-386 formulation 2(1 tab, once) / Period 3: D326, D337, D013(3 tabs, once)
  Interventions: Drug: CKD-386 formulation 1; Drug: CKD-386 formulation 2; Drug: D326, D337 and D013
- Sequence 2 (Experimental): Period 1: CKD-386 formulation 1(1 tab, once) / Period 2: D326, D337, D013(3 tabs, once) / Period 3: CKD-386 formulation 2(1 tab, once)
  Interventions: Drug: CKD-386 formulation 1; Drug: CKD-386 formulation 2; Drug: D326, D337 and D013
- Sequence 3 (Experimental): Period 1: CKD-386 formulation 2(1 tab, once) / Period 2: D326, D337, D013(3 tabs, once) / Period 3: CKD-386 formulation 1(1 tab, once)
  Interventions: Drug: CKD-386 formulation 1; Drug: CKD-386 formulation 2; Drug: D326, D337 and D013
- Sequence 4 (Experimental): Period 1: CKD-386 formulation 2(1 tab, once) / Period 2: CKD-386 formulation 1(1 tab, once) / Period 3: D326, D337, D013
  Interventions: Drug: CKD-386 formulation 1; Drug: CKD-386 formulation 2; Drug: D326, D337 and D013
- Sequence 5 (Experimental): Period 1: D326, D337, D013(3 tabs, once) / Period 2: CKD-386 formulation 1(1 tab, once) / Period 3: CKD-386 formulation 2(1 tab, once)
  Interventions: Drug: CKD-386 formulation 1; Drug: CKD-386 formulation 2; Drug: D326, D337 and D013
- Sequence 6 (Experimental): Period 1: D326, D337, D013 (3 tabs, once)/ Period 2: CKD-386 formulation 2(1 tab, once) / Period 3: CKD-386 formulation 1(1 tab, once)
  Interventions: Drug: CKD-386 formulation 1; Drug: CKD-386 formulation 2; Drug: D326, D337 and D013

INTERVENTIONS:
Drug: CKD-386 formulation 1 — A single oral dose of 1 tablet under fasting conditions for each period
  Other Names: CKD-386 Test 1
Drug: CKD-386 formulation 2 — A single oral dose of 1 tablet under fasting conditions for each period
  Other Names: CKD-386 Test 2
Drug: D326, D337 and D013 — A single oral dose of 3 tablets(D326, D337 and D013) under fasting conditions for each period
  Other Names: CKD-386 Reference

SUMMARY:
a study to investigate the pharmacokinetic characteristics and safety/tolerability according to formulations of CKD-386 in healthy male volunteers

DETAILED DESCRIPTION:
A sequence-randomized, open-label, 3-way crossover, single oral dose clinical trial to investigate the pharmacokinetic characteristics and safety/tolerability according to formulations of CKD-386 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between ≥20 and ≤45 years old
2. Weight ≥ 50 kg, with calculated body mass index(BMI) of ≥ 18.5 and ≤ 27.0 kg/m2
3. Those who have no congenital chronic disease or chronic disease requiring treatment and who have no pathological symptoms or findings
4. Those who are judged to be eligible for clinical trials based on laboratory and ECG results during screening tests
5. Those who voluntarily decide to participate and agree to comply with the cautions after hearing and fully understanding the detailed description of this clinical trial

Exclusion Criteria:

1. History of presence of hepatobiliary, renal, cardiovascular, endocrine, respiratory, gastrointestinal, hematological, neurologic, psychiatric or musculoskeletal disorders affecting absorption, distribution, metabolism and excretion of the drug
2. Genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
3. Those who are deemed unfit by the investigators to participate in the clinical trial for other reasons including the results of laboratory tests

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
AUC0-t of each main component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 or D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  AUC0-t: Area under the concentration-time curve from time zero to time
Cmax of each main component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 or D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf each main component or the metabolite of the component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~D3, Day15~D17, Day29~31
  AUCinf: Area under the concentration-time curve from zero up to ∞
Tmax of each main component or the metabolite of the component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  Tmax: Time to maximum plasma concentration
t1/2 of each main component or the metabolite of the component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  t1/2: Terminal elimination half-life
CL/F of each main component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  CL/F: Apparent total body clearance of the drug
Vd/F of each main component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  Vd/F: Apparent volume of distribution
AUC0-t of the metabolite of each component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  AUC0-t: Area under the concentration-time curve from time zero to time
Cmax of the metabolite of each component after single dose of CKD-386 formulation 1, CKD-386 formulation 2 and D326, D337, D013 | 0(predose)~72 hour at Day1~Day3, Day15~Day17, Day29~Day31
  Cmax: Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Dongseong Shin, M.D, Ph.D, Principal Investigator — Clinical Trials Center, Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No